CLINICAL TRIAL: NCT02834897
Title: Performance Evaluation of System EOS Imaging in Pelvimetry Versus Pelvi-scanner
Acronym: PELVI-EOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2014/236
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2016-07

CONDITIONS: Radiation; Obstetric Labor Complications; Pregnancy Complications
Keywords: EOS imagery
MeSH Terms: conditions — Obstetric Labor Complications; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EOS and CT Exam (Experimental): EOS and CT Examen for pregnant women in the 8th month of pregnancy
  Interventions: Radiation: EOS and CT Exam

INTERVENTIONS:
Radiation: EOS and CT Exam — EOS and CT Examen for pregnant women in the 8th month of pregnancy

SUMMARY:
The purpose of this study and demonstrate the reliability of EOS imaging system in the measurement of internal diameters of obstetrical pelvis versus "Goldstandard current "that is the pelviscanner.

ELIGIBILITY:
Inclusion Criteria:

* pelviscanner indication in women

Exclusion Criteria:

* In the disqualification of another study or under the "national register of volunteers."

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02-12 (Actual); Study Completion 2016-02-12 (Actual)

PRIMARY OUTCOMES:
Measurement reliability index Magnin with EOS cab relative to the CT measurements | one months

CONTACTS AND LOCATIONS:
Overall Officials: sebastien AUBRY, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHRU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No